CLINICAL TRIAL: NCT05448404
Title: A Head-to-head Comparative Study of 18F-PSMA-1007 PET/CT and 18F-FDG PET/CT Imaging in Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Xuena Li, Director, First Hospital of China Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 37587411
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Prostate specific membrane antigen; fluorodeoxyglucose; positron emission tomography/Computed Tomography
MeSH Terms: conditions — Multiple Myeloma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: 18F-PSMA-1007 PET/CT and 18F-FDG PET/CT Imaging completed within one week in the same patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PSMA-1007 and 18F-FDG PET/CT scan (Experimental): Patients of multiple myeloma PET/CT imaging: Within one week each patient underwent a PET/CT scan 60-min after intravenous administration of 18F-PSMA-1007 and 18F-FDG, respectively.
  Interventions: Drug: 18F-PSMA-1007; Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-PSMA-1007 — Intravenous injection of dosage of 222-370MBq(6-10mCi) 18F-PSMA-1007.
  Other Names: 18F-PSMA-1007 injection
Drug: 18F-FDG — Intravenous injection of dosage of 222-370MBq(6-10mCi) 18F-FDG.
  Other Names: 18F-FDG injection

SUMMARY:
Multiple myeloma (MM) is the second most common hematological malignancy and is still incurable. Positron emission tomography/computed tomography (PET/CT) has been used to diagnose, assess treatment response, and predict prognosis in MM. 18F-fluorodeoxyglucose (FDG) is the most widely used radiotracer, but there is heterogeneous uptake in MM, that is, uptake is negative in some myeloma cells. There are currently reports of cases with strong uptake of prostate-specific membrane antigen (PSMA) PET/CT in MM. Therefore, this preliminary study was designed to compare the imaging results of 18F-PSMA-1007 PET/CT and 18F-FDG PET/CT, and to evaluate the additional value of 18F-PSMA-1007 PET/CT to 18F-FDG PET/CT in MM.

DETAILED DESCRIPTION:
18F-fluorodeoxyglucose (FDG) PET/CT can identify bone lesions, assess disease burden, and detect extramedullary lesions in multiple myeloma(MM), but due to MM is a complex and heterogeneous disease , 18F-FDG PET/CT has heterogeneous uptake in MM bone lesions, resulting in false negative results in the diagnosis of MM bone disease, then affecting the diagnosis, staging and evaluation of the response to treatment of MM. Prostate-specific membrane antigen (PSMA) is a specific membrane-bound glycoprotein, recently high uptake in PSMA PET/CT in MM bone lesions has been published in case reports, thus PSMA PET CT imaging may have potential value for multiple myeloma. There are no head-to-head studies comparing 18F-PSMA-1007 PET/CT with 18F-FDG PET/CT in multiple myeloma. Therefore, this study intends to compare the detection rate of lesions by 18F-PSMA-1007 PET/CT and 18F-FDG PET/CT in MM , and to evaluate the additional value of 18F-PSMA-1007 PET/CT to 18F-FDG PET/CT in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* confirmed untreated or relapsed multiple myeloma patients;
* 18F-PSMA-1007 and 18F-FDG PET/CT within one week;
* signed written consent;
* no combined other Malignant tumors.

Exclusion Criteria:

* suffered from arthritis or combined with other malignant tumors;
* received myeloma-related therapy within 3 months before PET/CT imaging
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
number of myeloma lesions | through study completion, an average of 1 year
  comparing the number of myeloma lesions detected by 18F-PSMA-1007 and 18F-FDG PET

SECONDARY OUTCOMES:
standardized uptake value (SUV) of myeloma lesions | through study completion, an average of 1 year
  comparing the SUVmax of myeloma lesions derived from 18F-PSMA-1007 and 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided